CLINICAL TRIAL: NCT00605020
Title: Comparison of Efficacy and Safety of Insulin Detemir in Combination With Insulin Aspart and Biphasic Insulin Aspart 30 in Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety of Insulin Detemir in Combination With Insulin Aspart and Biphasic Insulin Aspart 30 in Type 2 Diabetes
Acronym: PreFER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1558
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir
  Other Names: Levemir
Drug: insulin aspart
Device: biphasic insulin aspart

SUMMARY:
This trial is conducted in Europe.

The aim of this trial is to investigate the efficacy and safety of an intensified treatment regimen with preprandial insulin aspart and insulin detemir once or twice daily to a more convenient regimen with biphasic insulin aspart 30 twice daily on blood glucose control in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Duration of type 2 diabetes for at least 6 months since diagnosis
* Current treatment with one or two oral antidiabetic drugs for at least 3 months or with one or two oral antidiabetic drugs, given for at least 3 months in combination with intermediate or long-acting insulin/insulin analogue once daily
* BMI below 40 kg/m2
* HbA1c between 7-12%
* Able and willing to perform self-monitoring of capillary blood glucose

Exclusion Criteria:

* Current antidiabetic treatment with combination of three or more oral antidiabetic drugs
* Previous treatment with short-acting human insulin, short-acting insulin analogue or biphasic insulin/insulin analogue within the last 6 months (7 days or less within the last 6 months is allowed)
* Known hypoglycaemia unawareness or recurrent major hypoglycaemia, as judged by the Investigator
* Known or suspected allergy to trial product or related products
* Pregnancy, breast-feeding, the intention of becoming pregnant or judged to be using inadequate contraceptive measures
* Receipt of any investigational drug within 4 weeks prior to this trial
* Previous participation in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 719 (Actual)
Dates: Start 2003-12-02 (Actual); Primary Completion 2005-03-03 (Actual); Study Completion 2005-03-03 (Actual)

PRIMARY OUTCOMES:
HbA1c | after 6 months of treatment

SECONDARY OUTCOMES:
Incidence of hypoglycaemic episodes
Adverse events
Difference of HbA1c change between the two groups | after 13 weeks of treatment
Fasting plasma glucose of treatment | after 13 and 26 weeks
Change in weight

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (109):
- Austria (3):
  - Novo Nordisk Investigational Site, Graz
  - Novo Nordisk Investigational Site, Linz
  - Novo Nordisk Investigational Site, Vienna
- Germany (101):
  - Novo Nordisk Investigational Site, Alsdorf
  - Novo Nordisk Investigational Site, Altenburg
  - Novo Nordisk Investigational Site, Altenkirchen
  - Novo Nordisk Investigational Site, Altenstadt
  - Novo Nordisk Investigational Site, Aschaffenburg
  - Novo Nordisk Investigational Site, Augsburg
  - Novo Nordisk Investigational Site, Bad Harzburg
  - Novo Nordisk Investigational Site, Bad Heilbrunn
  - Novo Nordisk Investigational Site, Bad Kreuznach
  - Novo Nordisk Investigational Site, Bad Lauterberg im Harz
  - Novo Nordisk Investigational Site, Bad Lippspringe
  - Novo Nordisk Investigational Site, Bad Mergentheim
  - Novo Nordisk Investigational Site, Bad Neuenahr-Ahrweiler
  - Novo Nordisk Investigational Site, Bad Oldesloe
  - Novo Nordisk Investigational Site, Bad Staffelstein
  - Novo Nordisk Investigational Site, Bensheim
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Bochum
  - Novo Nordisk Investigational Site, Damme
  - Novo Nordisk Investigational Site, Diez
  - Novo Nordisk Investigational Site, Dinslaken
  - Novo Nordisk Investigational Site, Dormagen
  - Novo Nordisk Investigational Site, Dortmund
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Duisburg
  - Novo Nordisk Investigational Site, Emmerich
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Flensburg
  - Novo Nordisk Investigational Site, Flörsheim
  - Novo Nordisk Investigational Site, Forchheim
  - Novo Nordisk Investigational Site, Frankfurt
  - Novo Nordisk Investigational Site, Freiburg im Breisgau
  - Novo Nordisk Investigational Site, Freital
  - Novo Nordisk Investigational Site, Gebhardshain
  - Novo Nordisk Investigational Site, Genthin
  - Novo Nordisk Investigational Site, Georgsmarienhütte
  - Novo Nordisk Investigational Site, Giessen
  - Novo Nordisk Investigational Site, Gotha
  - Novo Nordisk Investigational Site, Halle
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Hamelin
  - Novo Nordisk Investigational Site, Hanover
  - Novo Nordisk Investigational Site, Herne
  - Novo Nordisk Investigational Site, Herrenberg
  - Novo Nordisk Investigational Site, Hildesheim
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Hünxe
  - Novo Nordisk Investigational Site, Idar-Oberstein
  - Novo Nordisk Investigational Site, Jena
  - Novo Nordisk Investigational Site, Kaiserslautern
  - Novo Nordisk Investigational Site, Karlsruhe
  - Novo Nordisk Investigational Site, Krummennaab
  - Novo Nordisk Investigational Site, Künzing
  - Novo Nordisk Investigational Site, Landau
  - Novo Nordisk Investigational Site, Langen
  - Novo Nordisk Investigational Site, Lindenfels
  - Novo Nordisk Investigational Site, Lübeck
  - Novo Nordisk Investigational Site, Mainz
  - Novo Nordisk Investigational Site, Marburg
  - Novo Nordisk Investigational Site, Marktheidenfeld
  - Novo Nordisk Investigational Site, Meppen
  - Novo Nordisk Investigational Site, Mühlheim
  - Novo Nordisk Investigational Site, München
  - Novo Nordisk Investigational Site, Neumünster
  - Novo Nordisk Investigational Site, Neuwied
  - Novo Nordisk Investigational Site, Nittenau
  - Novo Nordisk Investigational Site, Northeim
  - Novo Nordisk Investigational Site, Oberhausen
  - Novo Nordisk Investigational Site, Oberndorf
  - Novo Nordisk Investigational Site, Oberursel
  - Novo Nordisk Investigational Site, Offenbach
  - Novo Nordisk Investigational Site, Osnabrück
  - Novo Nordisk Investigational Site, Pforzheim
  - Novo Nordisk Investigational Site, Pirna
  - Novo Nordisk Investigational Site, Regensburg
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Saaldorf
  - Novo Nordisk Investigational Site, Saarbrücken
  - Novo Nordisk Investigational Site, Saint Ingbert
  - Novo Nordisk Investigational Site, Sangerhausen
  - Novo Nordisk Investigational Site, Schaafheim
  - Novo Nordisk Investigational Site, Schkeuditz
  - Novo Nordisk Investigational Site, Schlüchtern
  - Novo Nordisk Investigational Site, Schwerin
  - Novo Nordisk Investigational Site, Schwerte
  - Novo Nordisk Investigational Site, Siegen
  - Novo Nordisk Investigational Site, Simmern
  - Novo Nordisk Investigational Site, Sinsheim
  - Novo Nordisk Investigational Site, Sögel
  - Novo Nordisk Investigational Site, Speyer
  - Novo Nordisk Investigational Site, Stuttgart
  - Novo Nordisk Investigational Site, Sulzbach-Rosenberg
  - Novo Nordisk Investigational Site, Trier
  - Novo Nordisk Investigational Site, Tübingen
  - Novo Nordisk Investigational Site, Völklingen
  - Novo Nordisk Investigational Site, Wallerfing
  - Novo Nordisk Investigational Site, Wangen
  - Novo Nordisk Investigational Site, Warburg
  - Novo Nordisk Investigational Site, Wiesbaden
  - Novo Nordisk Investigational Site, Wilhelmshaven
  - Novo Nordisk Investigational Site, Würzburg
- Switzerland (5):
  - Novo Nordisk Investigational Site, Basel-Bruderholz
  - Novo Nordisk Investigational Site, Geneva
  - Novo Nordisk Investigational Site, Lugano
  - Novo Nordisk Investigational Site, Sankt Gallen
  - Novo Nordisk Investigational Site, Zurich

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com